CLINICAL TRIAL: NCT02600767
Title: Evaluating the Efficacy of Artemether-lumefantrine for Treatment of Plasmodium Falciparum Malaria in Cruzeiro do Sul, Acre, Brazil
Brief Title: Artemether-lumefantrine for Treatment of P. Falciparum Malaria in Brazil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Secretaria Estadual de Saúde do Acre (Other); Ministry of Health, Brazil (Other Government); Evandro Chagas National Institute of Infectious Disease (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC-CGH-2015-204
Record Dates: First submitted 2015-10-22; First posted 2015-11-09 (Estimated); Results first posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2015-10

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Intervention Model Description: Evaluation of the efficacy of artemether and lumefantrine for uncomplicated P. falciparum malaria.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Artemether-Lumefantrine (Other): Three days of standard treatment. This is a standard combination therapy for the treatment of P. falciparum malaria.
  Interventions: Drug: Artemether-lumefantrine combination

INTERVENTIONS:
Drug: Artemether-lumefantrine combination — This is the sole arm in this study and it is the use of the standard combination therapy for treatment of P. falciparum malaria.
  Other Names: Coartem

SUMMARY:
This is an in vivo evaluation of drug efficacy performed in Cruzeiro do Sul, in the state of Acre, Brazil. A total of 81 participants ≥5 years old with parasitological confirmation of P. falciparum monoinfection will be treated under supervision with artemether-lumefantrine for three days, with doses according to the Brazilian guidelines for malaria control. The clinical and parasitological parameters will be monitored for a 28-day follow-up period to evaluate the efficacy of the combination therapy. A blood sample will be collected on filter paper on the first day and on the day of suspected failure to try to differentiate the parasite genotypes using techniques based on polymerase chain reactions. The results of this efficacy evaluation on the drug combination will help the Brazilian Ministry of Health to evaluate the national policy for treatment of malaria caused by P. falciparum.

DETAILED DESCRIPTION:
This protocol uses the recommended World Health Organization (WHO) protocol for monitoring antimalarial efficacy. Patients with malaria will receive supervised therapy and will be monitored for 28 days to check for treatment response, both clinically and parasitologically. A total of 81 participants ≥5 years old with parasitological confirmation of P. falciparum monoinfection will be treated under supervision with artemether-lumefantrine for three days, with doses according to the Brazilian guidelines for malaria control. The clinical and parasitological parameters will be monitored for a 28-day follow-up period to evaluate the efficacy of the combination therapy. Patients will be asked to come back on Days 2, 3, 7, 14, 21 and 28 for clinical evaluation and blood tests using microscopy. A blood sample will be collected on filter paper on the first day and on the day of suspected failure to try to differentiate the parasite genotypes using techniques based on polymerase chain reactions, this will allow us to determine if the recurrent infection was reinfection or failure or recrudescence. Results of this evaluation will guide treatment policies in Brazil.

ELIGIBILITY:
Inclusion Criteria:

* >= 5 years
* body weight < 120kg
* documented fever (axillary temperature ≥37.5o C) or history of fever in the previous 48 hours in the absence of other obvious causes of fever, such as pneumonia, middle ear infection, etc.
* monoinfection by P. falciparum with parasitemia between 250 and 200,000 asexual parasites/µl, as determined by swab and thick peripheral blood smear microscopic exam
* patient or parent/caregiver able to comprehend and sign informed consent or permission form
* patients aged 7-17 years able to provide assent, patients aged 5-6 years do not require assent
* willingness to return to the clinic and/or accept home visits for regular check-ups during the 28-day follow-up period
* hemoglobin level ≥8 g/dl

Exclusion Criteria

* presence of malaria danger signs (inability to drink, vomiting (more than twice in the previous 24 hours), recent history of seizures (one or more in the previous 24 hours), altered level of consciousness, inability to sit or stand up); presence of signs of severe malaria (altered level of consciousness, psychomotor alteration, seizure, torpor and irreversible coma), severe anemia (hematocrit < 15% or clinical signs, hemoglobin <5 g/dl), renal failure (serum creatinine > 3 mg/dl or clinical signs), pulmonary edema, hypoglycemia (blood glucose < 40 mg/dl or clinical signs), shock (systolic blood pressure < 70 mmHg for adults; < 50 mmHg for children), spontaneous hemorrhage/disseminated intravascular coagulation, repeated generalized seizures, acidemia/acidosis (clinical signs), macroscopic hemoglobinuria, and jaundice.
* history of chronic or severe underlying diseases (e.g. heart, renal or liver diseases, HIV/AIDS, tuberculosis, malnourishment)
* history of hypersensitivity to AL
* current pregnancy (history of current pregnancy or positive pregnancy test)
* use of any antimalarial drug in the previous 30 days.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Macedo de Oliveira, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Hospital do Jurua, Cruzeiro do Sul, Brazil

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Artemether-Lumefantrine
Started | 79
Completed | 74
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Artemether-Lumefantrine
Number analyzed (Participants) | 79
Age, Continuous [Median (Full Range); unit: years] | 30 [5 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 79
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 79

OUTCOME MEASURES:

1. Primary Outcome: Absence of Malaria Parasites in Blood.
Description: Investigators will evaluate the percentage of patients who remain free of malaria parasites in the blood during the 28-day follow-up period.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Artemether-Lumefantrine
Number analyzed (Participants) | 74
Participants | 73

ADVERSE EVENTS:
Arm/Group | Artemether-Lumefantrine
Serious Adverse Events (participants affected / at risk) | 0/79
Other Adverse Events (participants affected / at risk) | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No